CLINICAL TRIAL: NCT06890273
Title: Prospective NIS to Generate Real-World-Data on Effectiveness and Safety of First-line Therapy With Chemotherapy Combined With Durvalumab Followed by Maintenance Therapy With Durvalumab or Durvalumab + Olaparib in Endometrial Cancer
Brief Title: NIS to Examine the Effectiveness and Safety of Durvalumab and Olaparib in Patients With Endometrial Cancer (DUOLife)
Acronym: DUOLife
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: North-Eastern German Society of Gynecological Oncology (NOGGO e.V.) (Unknown)
Responsible Party: Sponsor
Other Study IDs: D9311R00001
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
Keywords: Durvalumab; Olaparib; Primary advanced endometrial cancer (1L); FIGO III or IV; Recurrent endometrial cancer (1L); dMMR; pMMR; Real-World Evidence; Patient-Reported Outcome
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DNA mismatch repair deficient (dMMR): Patients with primary advanced or recurrent endometrial cancer receiving 1L regimens of CPD with prior tested dMMR status. Following the SmPC patients of this cohort will receive durvalumab in the maintenance phase if they achieved and maintained disease control, i.e., complete response (CR), partial response (PR), or stable disease (SD) with CPD during the chemotherapy phase.
- DNA mismatch repair proficient (pMMR): Patients with primary advanced or recurrent endometrial cancer receiving 1L regimens of CPD with prior tested pMMR status. Following the SmPC patients of this cohort will receive durvalumab and olaparib in the maintenance phase if they achieved and maintained disease control i.e., CR, PR, or SD with CPD during the chemotherapy phase.

SUMMARY:
This is a German multi-center, prospective, non-interventional study (NIS) to collect real-world clinical and patient-reported outcome (PRO) data in patients with primary advanced (FIGO stage III or IV) or recurrent endometrial cancer (EC) receiving first-line (1L) regimens with Carboplatin/Paclitaxel/Durvalumab (CPD) followed by maintenance therapy with durvalumab or durvalumab and olaparib in line with the applicable european summary of product characteristics (SmPC).

DETAILED DESCRIPTION:
This is a multi-center, prospective, non-interventional study (NIS) to collect real-world clinical and PRO data in patients with primary advanced (FIGO stage III or IV) or recurrent EC receiving 1L CPD followed by maintenance therapy with durvalumab (DNA mismatch repair deficient; dMMR cohort) or durvalumab and olaparib (DNA mismatch repair proficient, pMMR cohort) in accordance with the applicable SmPC within routine clinical practice. Following surgery and/or radiation (if applicable) the decision to initiate 1L CPD followed by durvalumab or durvalumab and olaparib is made in a shared decision between the patient and the treating physician as part of routine care outside of and independent of this study.

The aim of the NIS is to describe the outcomes including effectiveness, safety and PRO of patients with primary advanced and recurrent EC treated with the two approved 1L regimens of CPD followed by durvalumab maintenance and CPD followed by durvalumab and olaparib maintenance in Germany. The study also aims to better understand characteristics of patients with primary advanced or recurrent EC that benefit from maintenance therapy with durvalumab or durvalumab and olaparib.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years at the time of screening.
* Patient has pathologically documented:
* Primary advanced (FIGO III and IV) epithelial EC OR
* Recurrent disease that is unlikely to be cured and where the multidisciplinary tumor board decision is systemic therapy. Carcinosarcomas are allowed,
* Patient is intended or initiated to receive 1L CPD followed by maintenance therapy with durvalumab (dMMR cohort) or with durvalumab and olaparib (pMMR cohort) according to the SmPC of IMFINZI® and Lynparza®* prior to enrollment. Recruitment of patients that already started and may have received up to 2 cycles of CPD is allowed but will be capped to 25% of the study population.
* Patient is eligible for treatment with durvalumab and/or olaparib as specified in the IMFINZI® and Lynparza® SmPC. The prescription of the medicinal product is clearly separated from the decision to include the patient in the study.
* MMR-testing results of the patient's tumor are known.
* Patient is willing and able to complete PRO questionnaires.
* Patient can read and understand German, English, Arab, Russian or Turkish.
* Signed written informed consent.

Exclusion Criteria:

* Patient has already received ≥2 cycles of 1L CPD
* Known hypersensitivity to carboplatin, paclitaxel, durvalumab and/or olaparib or any of the excipients of the drug.
* Pregnancy or breast-feeding.
* Unable to swallow orally administered medication.
* Current or planned participation in an interventional clinical trial.
* Current or planned systemic treatment of any tumor other than primary advanced or recurrent EC.
* Patient has pathologically documented sarcoma

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients with documented primary advanced (FIGO stage III or IV) or recurrent EC of epithelial histology (excluding sarcomas) who are eligible for first-line therapy with CPD followed by durvalumab or durvalumab and olaparib in line with the applicable SmPC within routine clinical practice will be recruited in Germany. The study allows recruitment of patients that already started and may have received up to 2 cycles of CPD. Inclusion of patients having started CPD will be capped to 25% of the study population. Testing results for MMR status of the patients' tumor must be available. Patients must be willing and able to report PROs. Eligible patients will be included into the study after and independently of the treating physician's treatment and diagnostic decisions.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Real-world Time To Next Treatment (rwTTNT) | At 12 months
  rwTTNT is defined as time from start of 1L CPD until the first dose of next systemic therapy or the start of any other next anticancer therapy or death from any cause.
  The measure of interest is the landmark at 12 months of time to first next therapy or death (rwTTNT).

SECONDARY OUTCOMES:
Real-world Progression-free Survival (rwPFS) | At 12 months
  rwPFS is defined as time from start of 1L CPD until progression or death from any cause.
  The measure of interest is the landmark at 12 months of progression-free survival (rwPFS).
Time to deterioration in health-related quality of life (HRQoL) based on EORTC QLQ-C30 questionnaire compared to baseline over time | Baseline to first clinically meaningful deterioration, up to 42 months
  The European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30), is a validated 30-item self-administered core questionnaire designed to assess HRQoL, functioning, and symptoms in all cancer patients or survivors.
  Time to deterioration is defined as time from baseline (defined as day 1 of cycle 1 before first application of maintenance therapy) to the date of the first clinically meaningful deterioration i.e. a decrease by ≥10 points for the functional scales and an increase by ≥ 10 points for the symptom scales or death in:
  * Physical functioning score
  * Role functioning score
Time to deterioration in HRQoL based on EORTC QLQ-EN24 questionnaire compared to baseline over time | Baseline to first clinically meaningful deterioration, up to 42 months
  The Endometrial Cancer Module EORTC QLQ-EN24, is a validated disease-specific extension to the EORTC QLQ-C30 designed to assess disease and treatment specific aspects of the QoLof patients with all stages of EC. The module consists of 24 questions grouped into 13 scales.
  Time to deterioration is defined as time from baseline (defined as day 1 of cycle 1 before first application of maintenance therapy) to the date of the first clinically meaningful deterioration i.e. a decrease by ≥10 points for the functional scales and an increase by ≥ 10 points for the symptom scales or death in:
  * Back/pelvic pain
  * Gastrointestinal (GI) symptoms
  * Urological symptoms
Treatment duration of maintenance therapy | From first dose of maintenance therapy up to 42 months
  Time from the first dose of maintenance therapy with durvalumab or durvalumab+olaparib to the last dose of durvalumab or olaparib, whatever is last, including number and duration of treatment interruptions.

OTHER OUTCOMES:
Safety: Collection of Adverse Events (AE) | During routine visits up to 42 months
  Safety evaluated based on type of Adverse Event (AE), intensity, causal relationship to treatment, duration, handling, outcome, and seriousness.
Change in timed up and go test (TUG) | Baseline up to 42 months
  The Timed up and go test (TUG) is a reliable and validated measure of functional mobility that can be used to assess frailty and functional impairment and to predict the risk of postoperative complications. The TUG records the time it takes a patient to get up from an armchair, walk 3 meters, turn around, walk back, and sit down again. Aids such as walking aids are permitted but help from other people is not.
  TUG should be assesd at every routine visit.
Change in EORTC QLQ-C30 | Baseline up to 42 months
  Changes of patient-reported outcomes (PROs) based on the European Organisation for Research and Treatment of Cancer Quality of Life - Core Questionnaire 30 (EORTC QLQ-C30) questionnaire from baseline (defined as day 1 of cycle 1 before application of first dose of maintenance therapy) over time in:
  * Physical functioning score of EORTC QLQC30
  * Role functioning score of the EORTC QLQ-C30
  * Global health status/quality of life (QoL) score of the EORTC QLQ-C30
  * All other functioning and symptom subscale scores of the EORTC QLQ-C30.

CONTACTS AND LOCATIONS:
Locations (15):
- Germany (15):
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Borna
  - Research Site, Bottrop
  - Research Site, Brandenburg
  - Research Site, Dessau
  - Research Site, Ebersberg
  - Research Site, Gütersloh
  - Research Site, Landshut
  - Research Site, Leipzig
  - Research Site, Lüneburg
  - Research Site, Mainz
  - Research Site, Plauen
  - Research Site, Unna
  - Research Site, Worms

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved, AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://vivli.org/